CLINICAL TRIAL: NCT07198035
Title: A PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD STUDY IN HEALTHY PARTICIPANTS TO INVESTIGATE THE EFFECT OF CARBAMAZEPINE ON PF-07248144 PHARMACOKINETICS
Brief Title: A Study to Learn if Multiple Doses of the Study Medicine Called Carbamazepine Changes How the Body Processes the Other Study Medicine PF-07248144
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: C4551007; 2025-522331-34-00 (Registry Identifier: CTIS (EU))
Record Dates: First submitted 2025-09-25; First posted 2025-09-30 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Healthy Adults
MeSH Terms: interventions — Carbamazepine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- PF-07248144 with and without Carbamazepine (Experimental): PF-07248144 administered as a single dose in Period 1 on Day 1 and in Period 2 on Day 14.
  Carbamazepine administered once a day for Day 1 through 3, then twice a day for Day 4 through 7, and then three times daily for Day 8 through 20 in Period 2
  Interventions: Drug: PF-07248144; Drug: Carbamazepine

INTERVENTIONS:
Drug: PF-07248144 — Participants will receive a single dose of PF-07248144 by mouth in Period 1 on Day 1 and Period 2 on Day 14, with a washout period of at least 14 days between two doses of PF-07248144
Drug: Carbamazepine — Participants will receive Carbamazepine by mouth once a day for Day 1 through 3, then twice a day for Day 4 through 7, and then three times daily for Day 8 through 20 in Period 2.
  Other Names: Tegretol

SUMMARY:
The purpose of the study is to learn how the study medicine called carbamazepine changes how the body processes the other study medicine called PF-07248144. The study will also look at the safety, tolerability, and how PF-07248144 is changed and removed from the body after taking PF-07248144 alone compared to when it is taken with carbamazepine.

Carbamazepine can change how your body processes some medications so it may change the body's processing of PF-07248144. Multiple blood samples will be collected up to 8 days after each dose of PF-07248144 to determine how much PF-07248144 is in the blood at different times. This will help characterize the pharmacokinetics (pharmacokinetics helps us understand how the drug is changed and eliminated from your body after you take it) of PF-07248144 alone and when taken with carbamazepine.

ELIGIBILITY:
Inclusion

* Females of nonchildbearing potential and males, inclusive, at screening who are able to provide consent and are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, vital signs, and 12-lead electrocardiogram (ECG)s.
* Body mass index (BMI) of 16-32 kg/m2; and a total body weight >45 kg (99 lb).

Exclusion

* Participants shown to carry or be positive for human leukocyte antigen (HLA)-B*1502 and/or HLA-A*3101 (genotyping alleles/markers related with carbamazepine-associated Stevens-Johnson syndrome (SJS) or toxic epidermal necrolysis [TEN]).
* Any medical or psychiatric condition including any active suicidal ideation in the past year or suicidal behavior in the past 5 years or laboratory abnormality that may increase the risk of study participation or, in the investigator's judgment, make the participant inappropriate for the study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 14 days or 5 half-lives (whichever is longer) prior to the first dose of study intervention.
* Additionally, current use or anticipated need for food or drugs that are known moderate or strong inducers or inhibitors of CYP2C9 or CYP3A4, including their administration within 14 days or 5 half-lives of the strong inducers or inhibitors of CYP2C9 or CYP3A4, whichever is longer, prior to first dose of study intervention, during the treatment period, and within 10 days after the last dose of PF-07248144.
* Pregnant female participants; breastfeeding female participants; individual(s) of childbearing potential (IOCBPs); fertile male participants who are unwilling or unable to use highly effective methods of contraception as outlined in this protocol for the duration of the study and for at least 103 days after the last dose of study intervention.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-09-18 (Actual); Primary Completion 2025-12-19 (Estimated); Study Completion 2025-12-26 (Estimated)

PRIMARY OUTCOMES:
Maximum Observed Plasma Concentration (Cmax) Period 1 | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120 and 168 hours post-dose
Cmax Period 2 | Day 14: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120 and 168 hours post-dose
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) Period 1 | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120 and 168 hours post-dose
AUCinf Period 2 | Day 14: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120 and 168 hours post-dose
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast). Period 1. To be used as the primary endpoint if AUCinf cannot be reliably estimated | 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120 and 168 hours post-dose
AUClast. Period 2. To be used as the primary endpoint if AUCinf cannot be reliably estimated | Day 14: 0 (pre-dose), 0.5, 1, 2, 3, 4, 6, 8, 12, 24, 36, 48, 72, 120 and 168 hours post-dose

SECONDARY OUTCOMES:
Number of Treatment-Emergent Treatment-Related AEs by Severity | From Day 1 of dosing up to 35 days after last of study intervention (maximum up to 55 days)
Number of Participants With Laboratory Test Abnormalities | From Day 1 of dosing up to 35 days after last of study intervention (maximum up to 55 days)
Number of Participants With Clinically Significant Physical Examination Abnormalities | From Day 1 of dosing up to 35 days after last of study intervention (maximum up to 55 days)
Number of Participants With Vital Signs Values Meeting Categorical Summarization Criteria | From Day 1 of dosing up to 35 days after last of study intervention (maximum up to 55 days)
Number of Participants With Clinically Significant Changes From Baseline in 12-Lead Electrocardiogram (ECG) Parameters | From Day 1 of dosing up to 35 days after last of study intervention (maximum up to 55 days)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Clinical Research Unit - Brussels, Brussels, Other, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=C4551007